CLINICAL TRIAL: NCT00070837
Title: A Phase 1/2 Dose Escalation Trial of Multiple Doses of MLN2704 (DM1 Conjugated Monoclonal Antibody MLN591) in Subjects With Metastatic Androgen-Independent Prostate Cancer
Brief Title: MLN2704 in Subjects With Metastatic Androgen-Independent Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M59102-051; NCT00074347 (obsolete NCT alias)
Expanded Access: Available
Record Dates: First submitted 2003-10-08; First posted 2003-10-13 (Estimated); Last update posted 2007-07-13 (Estimated); Status verified 2007-07

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms

INTERVENTIONS:
Drug: MLN2704 (DM1 conjugated monoclonal antibody MLN591)

SUMMARY:
The purpose of the study is to determine the highest dose of MLN2704 that can be given multiple times safely to patients with prostate cancer, and to identify any side effects associated with taking the drug. This study will also evaluate how MLN2704 is taken up, broken down and eliminated by the body.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis (recent or remote) of prostate adenocarcinoma
* Radiographic evidence (recent or remote) of metastatic prostate adenocarcinoma
* 18 years of age or older
* Progressive prostate cancer as defined by the presence of one or more of the following despite castrate levels of testosterone (testosterone <50 ng/dL):

  1. Progressive tumor lesions (changes in the size of lymph nodes or parenchymal masses on physical examination or X-ray and CT scan or MRI)
  2. Progressive bone metastasis (presence of new lesion(s) on a bone scan)
  3. Progressive PSA levels (as defined in Section 3.6.1)
* Subjects who have received an anti-androgen must have shown progression of disease following discontinuation of the anti-androgen
* Subjects must remain on luteinizing hormone-releasing hormone (LHRH) analog therapy for the duration of the trial unless surgically castrate
* Agree to use an effective barrier method of contraception.

Exclusion criteria:

* Testosterone >50 ng/dL
* Use of corticosteroids and/or adrenal hormone inhibitors within 4 weeks of dosing
* Use of PC-SPES within 4 weeks of dosing
* Prior cytotoxic chemotherapy and/or radiation therapy within 6 weeks of dosing
* Use of anti-androgen therapy (eg, flutamide, bicalutamide, nilutamide) within 6 weeks of dosing
* Prior monoclonal antibody administration, including Prostascint®
* Peripheral neuropathy of > Grade 2, as defined by the NCI Common Toxicity Criteria for Adverse Events (NCI CTCAE)
* History of CNS metastasis, including incompletely treated epidural disease
* History of Hepatitis B or C
* History of seizure disorder requiring active treatment and/or stroke
* History of HIV infection
* Platelet count <100,000/mm3
* Absolute neutrophil count (ANC) <1,500/mm3
* Hematocrit <27 percent
* Abnormal coagulation profile (elevated PT, and/or INR, PTT)
* Serum creatinine >2.0 mg/dL, or creatinine clearance <60 mL/min if serum creatinine >2.0 mg/dL
* AST or ALT >1.5 x ULN
* Bilirubin (total) >1.25 x ULN
* Serum calcium >12.5 mg/dL
* Active serious infection not controlled by antibiotics
* Active angina pectoris or NY Heart Association Class III-IV heart disease
* Karnofsky Performance Status <60%
* Life expectancy <6 months
* Other serious illness(es) involving the cardiac, respiratory, CNS, renal, hepatic or hematological organ systems that might preclude completion of this study or interfere with determination of causality of any adverse effects experienced in this study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46
Dates: Start 2003-10; Study Completion 2004-10

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Weill Medical College of Cornell University/ New York Presbyterian Hospital, New York, New York
  - Duke University Medical Center, Box 3532, Durham, North Carolina
  - Cleveland Clinic, Taussig Cancer Center, Cleveland, Ohio